CLINICAL TRIAL: NCT00743041
Title: The Effect of EFT (Emotional Freedom Techniques) on Psychological States in a Veterans Population: A Randomized Controlled Trial
Brief Title: The Effect of EFT on Psychological States in a Veterans Population
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Soul Medicine Institute (Other)
Responsible Party: Dawson Church, Executive Director, Soul Medicine Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: SMI-PTSD-82508
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: PTSD, EFT, depression, anxiety, telephone
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Standard of Care plus EFT (Emotional Freedom Techniques)
  Interventions: Behavioral: Emotional Freedom Techniques (EFT)
- 2 (No Intervention): Standard of Care (SOC)

INTERVENTIONS:
Behavioral: Emotional Freedom Techniques (EFT) — EFT is an exposure therapy with a cognitive component, consisting of recall of a trauma along with a statement of self-acceptance, in combination with touching or tapping on a series of stress reduction points on the body
  Other Names: EFT Emotional Freedom Technique
  Arms: 1

SUMMARY:
A need exists to find fast yet effective treatment protocols for the large number of US military service personnel coming back from Iraq with post traumatic stress disorder (PTSD), and a variety of co-occurring psychological problems. EFT (Emotional Freedom Techniques) has demonstrated promise as a PTSD treatment in pilot studies. This study examines the effects of six sessions of EFT coaching on veterans who score at or above the military cutoff point for PSTD. Subjects are also assessed for conditions that often accompany PTSD, such as depression and anxiety. Changes pain, cravings, and physical symptoms are also measured. Assessments are made after six sessions are complete, and again after three and six months.

DETAILED DESCRIPTION:
A need exists to find fast yet effective treatment protocols for the large number of US military service personnel coming back from Iraq with post traumatic stress disorder (PTSD), and a variety of co-occurring psychological problems. This study examines the effects of six sessions of EFT coaching on a veterans population. The sample will recruited from clients of practitioners who are coaching veterans. Participants will be assessed for PTSD and other psychological conditions such as anxiety and depression. Evaluations will be made using well-validated instruments, the SA-45 (Symptom Assessment 45) and the PCL-M (Posttraumatic Stress Disorder Checklist - Military). Those meeting the military's criterion for a PTSD-positive assessment on the PCL-M will be randomized into two groups. A wait list control group continues to receive Standard of Care (SOC) from their current healthcare provider. The experimental group receives SOC plus EFT coaching. A baseline measurement is obtained approximately thirty days in advance of coaching, when subjects apply to participate in the study, and again immediately before coaching begins. Participants are assessed after three sessions and six sessions, to determine symptom changes at these milestones. Followup assessments occur three months and six months post-coaching. Pain levels, alcohol use, recreational drug use, and prescription drug dosages are also tracked, in order to determine any correlation between participant characteristics and psychological symptom change. Data will also be analyzed to determine if there are outcome differences between participants receiving EFT from life coaches, and those whose EFT coaching is delivered by licensed psychologists or social workers.

ELIGIBILITY:
Inclusion Criteria:

* Military Service
* Score of 50 or more on the PCL-M (PTSD Checklist-Military)
* The ability to follow instructions and complete written forms
* Under the care of a primary care provider

Exclusion Criteria:

* A score of 3 or more on questions 34 and 35 of the SA-45

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Scores on the PCL-M (PTSD Symptom Checklist-Military) | One Month Before, At Start, After 3 and 6 Sessions, After 3 and 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Dawson Church, PhD, Principal Investigator — Soul Medicine Institute
Locations (1):
- Soul Medicine Institute, Santa Rosa, California, United States

REFERENCES:
- [Background] Geronilla, L., Minewiser, L., Mollon, P., McWilliams, M., & Clond, M. (2016). EFT (Emotional Freedom Techniques) remediates PTSD and psychological symptoms in veterans: A randomized controlled replication trial. Energy Psychology: Theory, Research, and Treatment, 8(2), 29-41. doi:10.9769/EPJ.2016.8.2.LG
- See also: National Institute for Integrative Healthcare — http://www.NIIH.org